CLINICAL TRIAL: NCT05151575
Title: The Effects of Walking on Frailty, Cognitive Function and Quality of Life Among Inactive Older Adults in Saudi Arabia: A Randomized Control Trial by Comparing Supervised Group-based Intervention and Non-supervised Individual-based Intervention
Brief Title: Supervised Group-based Walking Intervention Among Inactive Older Adults in Saudi Arabia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 24_PH_in_Sport_Chung
Record Dates: First submitted 2021-11-08; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Physical Activity
Keywords: Ageing; Older Adults; Physical activity; Group-based intervention; Quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group-based walking intervention with professional trainer's supervision (Experimental): Participants will conduct the intervention in groups under the supervision of a professional fitness trainer.
  Interventions: Behavioral: supervised group-based walking and non-supervised individual-based walking interventions
- individual-based walking intervention without professional trainer supervision (Active Comparator): Participants will conduct the intervention individually, without the supervision of a professional fitness trainer
  Interventions: Behavioral: supervised group-based walking and non-supervised individual-based walking interventions
- control group (No Intervention): No intervention will be given to the control group.

INTERVENTIONS:
Behavioral: supervised group-based walking and non-supervised individual-based walking interventions — Group exercise interventions tended to be systematic and supervised by professionals. The current intervention is proposing to conduct a randomized control trial that is not only examining the nature of walking on older adults' well-being but also involving the elements of group-based and professional supervision intervention, aiming at comparing with the individual-based intervention without professional supervision. Qualified professional fitness trainers (1 male and 1 female separately for male and female groups, respectively) will be involved in the group-based intervention programs in order to provide appropriate guidance and supervision to the participants. Whereas, the non-supervised individual-based intervention will be conducted by a research assistant (males and females) to ensure the attendance and general safety, but without providing professional advice or supervision.
  Arms: group-based walking intervention with professional trainer's supervision; individual-based walking intervention without professional trainer supervision

SUMMARY:
The purpose of the proposed study is to compare the effects of supervised group-based walking and non-supervised individual-based walking interventions on frailty, cognitive function and quality of life among inactive older adults in Saudi Arabia.

DETAILED DESCRIPTION:
Objectives

1. To compare the difference of effects between supervised group-based walking and non-supervised individual-based walking on the primary outcomes, including frailty, cognitive functions, and health-related quality of life among inactive older adults in Saudi Arabia.
2. To compare the difference of effects between supervised group-based walking and non-supervised individual-based walking on the secondary outcomes, including physical activity enjoyment, health parameters consisting of resting heart rate, resting blood pressure, and body composition, as well as walking performance among inactive older adults in Saudi Arabia.
3. To formulate guidelines for achieving an effective walking intervention for inactive older adults in Saudi Arabia.
4. To recommend the government of Saudi Arabia on guidelines and policies for promoting walking and active ageing among the older adults in the country.

ELIGIBILITY:
Inclusion Criteria:

* 60-70 years old
* capable of walking without assistive device
* healthy and live independently in communities
* being physically inactive

Exclusion Criteria:

* with cardiovascular or related diseases that prevent from intensive walking
* fail the PAR-Q screening or without physician's advice on readiness of participation in exercise training
* diagnosed with cognitive impairment

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Health-related quality of life at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The Short Form-36 (SF-36) is a widely used health survey questionnaire, especially for older adults to assess the health-related quality of life (HRQoL). The higher the scores mean a higher level of quality of life.
Change from baseline Frailty level at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  Physical Performance Test (PPT) is one of the tools which is used to assess the level of frailty. For our research we will use 9 item scale that includes 9 standardized tasks such as writing a sentence, simulated eating, turning 360 degrees, putting on and removing a jacket, lifting a book and putting it on a shelf, picking up a penny from the floor, a 50-foot walk test, and climbing stairs (scored as two items) (Reuben and Siu, 1990). The score range of each task is 0-4 and for 9 items it will be 36. A higher score indicates better performance (Villareal et al., 2017).
Change from baseline Cognitive function at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The Mini-mental state examination (MMSE) is the most commonly used method to measure the level of cognitive impairment, especially in older adults. The score of Mini-mental state examination is calculated on a scale of 0-30 where score 24 or above is usually considered as the normal cognitive status or no cognitive impairment of the individual. The overall scorings are Severe cognitive impairment (0-17), Mild cognitive impairment (18-23) and No cognitive impairment (24-30).

SECONDARY OUTCOMES:
Change from baseline Health parameters - Body Composition at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The walking effects on participants' health parameters, namely body composition, will be assessed. The body composition will be assessed by Tanita MC780U (Tanita Corporation, 2020), by which the percent body fat and lean body mass of participants will be recorded. The body mass index (BMI) using participants' heights and weights (measured by the RA) will also be recorded.
Change from baseline Health parameters - Resting Heart Rate at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The walking effects on participants' health parameters, namely resting heart rate, will be assessed. The wrist-worn Fitbit Charge 3 (Fitbit, Inc., 2020) will be used to record the resting heart rate of participants (also the heart rates during walking for reflecting the exercise intensity of the participants as well as the accumulated footsteps and the duration of the completed footsteps during each session of the intervention for performance analyses).
Change from baseline Health parameters - Resting Blood Pressure at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The walking effects on participants' health parameters, namely resting blood pressure, will be assessed. The resting blood pressure of the participants will be recorded by Lenus Automatic Blood Pressure Monitor DP65 (MDF Instruments USA, 2020).
Change from baseline Physical Activity Enjoyment at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The 8-item Physical Activity Enjoyment Scale (PACES; Chung & Leung, 2019) will be applied to measure the participants' level of enjoyment after engaging in walking intervention programs. The 8-item Physical Activity Enjoyment Scale is rated by a 7 bipolar rating, with items such as " I enjoy it." (one extreme) to " I dislike it."(the other extreme). In the scale, the negative items (i.e., 1, 4, 5, and 7) requires reverse coding, and the Higher PACES scores the greater levels of physical activity enjoyment demonstrated.
Change from baseline Walking Performance at 4 months and at 7 months | Time 1: Baseline; TIme 2 after the 16-week intervention; Time 3 12-weeks after the intervention
  The time for completing the targeted steps in targeted heart rate zones of each participant in each training session will be recorded for analysis of performance and improvement on walking. All the data will be recorded by the wrist-worn Fitbit Charge 3 (Fitbit, Inc., 2020) and retrieve from the computer after each training session.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Pak Kwong, Prof, Principal Investigator — Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong MYC, Karmakar P, Almarzooqi MA, Rhodes RE, Zhang CQ, Ou KL, Yanping D, Chung PK, Alghamdi NA. The effects of walking on frailty, cognitive function and quality of life among inactive older adults in Saudi Arabia: a study protocol of randomized control trial by comparing supervised group-based intervention and non-supervised individual-based intervention. BMC Geriatr. 2023 Sep 27;23(1):602. doi: 10.1186/s12877-023-04200-w. PMID 37759212